CLINICAL TRIAL: NCT06227819
Title: BVA-200 vs BVA-100 Validation Study
Status: Completed | Type: Observational
Sponsor: Daxor Corporation (Industry)
Collaborators: Stern Cardiovascular Foundation, Inc. (Industry); Oregon Health and Science University (Other)
Responsible Party: Sponsor
Other Study IDs: BVA-200 Validation
Record Dates: First submitted 2023-12-29; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Heart Failure; High Blood Pressure; High Cholesterol; Anemia; Diabetes; Thyroid Diseases; Kidney Diseases; Clotting Disorder; Trauma; Other Disease
Keywords: Blood volume; Point of care; Fluid management; Diagnostic
MeSH Terms: conditions — Heart Failure; Hypertension; Hypercholesterolemia; Anemia; Diabetes Mellitus; Thyroid Diseases; Kidney Diseases; Hemostatic Disorders; Wounds and Injuries; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: BVA-200 — Blood samples collected for measurement with the BVA-100 will also be tested with the BVA-200. The BVA-200 uses whole blood collection cartridges which allow for a precise amount of blood to be measured without the need to first centrifuge and then pipette plasma aliquots. A small amount of whole blood from each sample will be set aside for BVA-200 use, while the remainder of the blood sample is used for BVA-100 measurement. The BVA-200 device was developed with the support of the Department of Defense through Phase I (W81XWH19C0048) and Phase II (W81XWH20C0025) SBIR contracts.

SUMMARY:
The proposed study is a prospective, observational, investigator and patient blinded study comparing the results of blood volume measurement using the FDA-cleared Daxor BVA-100 device to the Daxor BVA-200 device. Data from this study may be pooled with data from studies with similar design conducted at other sites, for the purposes of an FDA medical device submission.

DETAILED DESCRIPTION:
Measurements of human blood volume will be made via the indicator dilution method, using gamma counter readings of the concentration of I-131 in a subject's blood sample taken after radio-iodinated Human Serum Albumin (HSA) has been injected into the bloodstream via venous access. Each subject receiving an injection will have five separate blood samples taken, which will be analyzed separately. Each of the five measurements will be conducted in duplicate with the BVA-100 instrument and the BVA-200 instrument. Sufficient blood will be withdrawn at each phlebotomy to permit such duplicate measurement.

Subjects will be enrolled who have been prescribed a blood volume procedure using the BVA-100, as a result either of their ordinary diagnostic care or of their participation in another study that uses blood volume measurement. Subjects will be adults under treatment for conditions normally associated with the need for volume assessment, such as Heart Failure, or scheduled to receive BVA-100 measurement as part of another study. An effort will be made to ensure a range of ages and a balance of the sexes.

Subjects will be enrolled and consented sequentially. The University of Tennessee Medical Center site will document any patient who is not enrolled in the study sequentially and the reason why or who declines enrollment. Demographics of patients not enrolled will be collected to permit identification of any trends in non-enrollment. We do not anticipate any sequential patient not being offered the opportunity to participate in order to assure that there is no bias in selection of patients ("all-comers").

ELIGIBILITY:
Inclusion Criteria:

1. Age: Over18 years;
2. Able and willing to provide informed written consent.
3. Subjects will be enrolled who have been prescribed a blood volume procedure using the BVA-100, as a result either of their ordinary diagnostic care or of their participation in another study that uses blood volume measurement. Subjects will be adults under treatment for conditions normally associated with the need for volume assessment, such as Heart Failure, or scheduled to receive BVA-100 measurement as part of another study.

Exclusion Criteria:

1. Pregnant women or nursing mothers.
2. Women of childbearing potential not using adequate birth control methods.
3. Known hypersensitivity to iodine or eggs.
4. Other clinical basis for precluding the use of radioactive materials.
5. Has previously been enrolled in, and completed, the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The proposed study will be open to any volunteer meeting the inclusion/exclusion criteria listed below. We intend to highlight differential analysis of clinical patients from exemplary disease states (such as congestive heart failure and chronic kidney disease), as well as other population characteristics such as age, sex, race, etc.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Establish equivalence of BVA-200 to BVA-100 | Approximately 6 months.
  Comparison of a sufficient number of indicator-dilution volume measurements between BVA-100 and BVA-200 devices to establish substantial equivalence.

SECONDARY OUTCOMES:
Establish equivalence of BVA-200 to BVA-100 in TBV, RCV, PV and ATR | Approximately 6 months.
  Comparison of a sufficient number of full 5-point time-zero blood volume measurements between BVA-100 and BVA-200 devices, to establish substantial equivalence, including measurement of:
  * Total Blood Volume (TBV)
  * Red Cell Volume (RCV)
  * Plasma Volume (PV)
  * Albumin transudation rate (ATR)
Filling consistency validation | Approximately 6 months.
  Validation of filling consistency of at least 100 whole blood quantitative collection cartridges, in at least 40 sets of 5 samples from the same patient
Usability | Approximately 6 months.
  Validation of the ability of personnel who are not laboratorians to understand the test procedures and perform the measurement after receiving training materials (which may be a combination of written instructions, video instructions, and individual instruction) in the use of the instrument. Usability is evaluated through a User Validation Survey consisting of yes or no questions, as well as questions answered on a scale of 1 (strongly disagree) to 5 (strongly agree), where 5 is the most favorable outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Feldschuh, Principal Investigator — Daxor Corporation
Locations (1):
- Daxor Corporation, Oak Ridge, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be made available to other researchers.